CLINICAL TRIAL: NCT04838496
Title: Neo-adjuvant FOLFOXIRI and Chemoradiotherapy for High Risk ("Ugly") Locally Advanced Rectal Cancer
Brief Title: Induction Chemotherapy for Locally Advanced Rectal Cancer
Acronym: MEND-IT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, J. W. A. Burger, Principal investigator, Catharina Ziekenhuis Eindhoven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL74465.100.20
Record Dates: First submitted 2021-04-02; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Rectal Cancer
Keywords: Locally advanced rectal cancer; Induction chemotherapy; Neoadjuvant chemotherapy; Chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — FOLFOXIRI protocol

STUDY DESIGN:
Intervention Model Description: This is a multicentre, single-arm, prospective phase 2 study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm study (Experimental): All patients will receive induction chemotherapy consisting of 4-6 cycles of FOLFOXIRI. Restaging will be performed after 4 cycles with a pelvic MRI and a thoraco-abdominal CT-scan. In case of stable or responsive disease, the remaining 2 cycles of FOLFOXIRI will be provided. In case of progressive, but still resectable disease, chemoradiation will be provided immediately, without the remaining 2 cycles of FOLFOXIRI. Restaging will be performed after chemoradiation. In case of resectable disease, surgery is performed.
  Interventions: Drug: FOLFOXIRI Protocol

INTERVENTIONS:
Drug: FOLFOXIRI Protocol — FOLFOXIRI consists of oxaliplatin, irinotecan, leucovorin and 5-fluorouracil and is administered every 2 weeks:
  Dosing:
  * Day 1: irinotecan 165 mg/m2 body-surface area (BSA) intravenously (IV), followed by oxaliplatin 85mg/m2 BSA IV in combination with leucovorin 400mg/m2 BSA, followed by:
  * Day 1-2: 3200 mg/m2 BSA of continuous 5-fluorouracil IV
  * Day 3-14: rest days.
  Both regimen are initially administered for four cycles. In case of responsive or stable disease, a 5th and 6th cycle of FOLFOXIRI will be administered.
  In case of unacceptable toxicity, the aforementioned dosages can be reduced or one or more chemotherapeutical agents can be omitted at discretion of the medical oncologist and will be noted in the patient's medical file. At discretion of the medical oncologist, a start dosage of 75% of the advised dosage could be considered in patients above 70 years of age.

SUMMARY:
Despite developments in the multidisciplinary treatment of patients with locally advanced rectal cancer (LARC), such as the introduction of total mesorectal excision (TME) by Heald et al. and the shift from adjuvant to neoadjuvant (chemo)radiotherapy ((C)RT), local and distant recurrence rates remain between 5-10% and 25-40% respectively. Several studies established tumour characteristics with particularly bad prognosis; it was demonstrated that the occurrence of mesorectal fascia involvement (MRF+), grade 4 extramural venous invasion (EMVI), tumour deposits (TD) and enlarged lateral lymph nodes (LLN) lead to high local and distant recurrence rates and decreased survival when compared with LARC without these particularly negative prognostic factors. This type of LARC is described as high risk LARC (hr-LARC). Achieving a resection with clear resection margins (R0) is an important prognostic factor for local (LR) and distant recurrence (DM) as well as survival. With the aim to further reduce the risk of recurrent rectal cancer, to diminish distant metastasis and to improve overall survival for patients with LARC, induction chemotherapy (ICT) became a growing area of research. The addition of ICT has the ability to induce more local tumour downstaging, possibly leading to resectability of previously unresectable tumours, more R0 resections and less extensive surgery. In the case of a complete clinical response, surgery may even be omitted. ICT may also have the potential to eradicate micrometastases. Hence, increased local downstaging and reducing distant metastatic spread may reduce LR and DM rates and improve survival and quality of life. In recent years, the use of ICT was investigated and showed promising results, but little is known about the addition of ICT in patients with high risk LARC. Since these patients have a particularly bad prognosis, both with regard to locoregional and distant failure, a more intensified neoadjuvant treatment with FOLFOXIRI is anticipated to improve short- and long term results.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* WHO performance score 0-1.
* Histopathologically confirmed rectal cancer.
* Lower border of the tumour located below the sigmoidal take-off as established on MRI of the pelvis.
* Confirmed high-risk locally advanced rectal cancer, meeting one of the following imaging based criteria:

  * Tumour invasion of mesorectal fascia (MRF+)
  * The presence of grade 4 extramural venous invasion (mrEMVI)
  * The presence of tumour deposits (TD)
  * The presence of Extramesorectal lymph nodes with a short-axis size > 7mm (LNN)
* Resectable disease as determined on magnetic resonance imaging (MRI) or deemed resectable disease after neoadjuvant treatment.

Expected gross incomplete resection with overt tumour remaining in the patient after resection, tumour invasion in the neuroforamina, encasement of the ischiadic nerve and invasion of the cortex from S3 and upwards are considered not resectable • Written informed consent.

Exclusion Criteria:

* Evidence of metastatic disease at the moment of inclusion or within six months prior to inclusion except for patients with enlarged iliac or inguinal lymph nodes and aspecific lung noduli.
* Homozygous DPD (Dihydropyrimidine dehydrogenase) deficiency.
* Any chemotherapy within the past 6 months.

  o Any contraindication for the planned systemic therapy (e.g. severe allergy, pregnancy, kidney dysfunction and thrombocytopenia), as determined by the medical oncologist.
* Radiotherapy in the pelvic area within the past 6 months.
* Any contraindication for the planned chemoradiotherapy (e.g. severe allergy to the chemotherapy agent or no possibility to receive radiotherapy), as determined by the medical oncologist and/or radiation oncologist.
* Any contraindication to undergo surgery, as determined by the surgeon and/or anaesthesiologist.
* Concurrent malignancies that interfere with the planned study treatment or the prognosis of the resected tumour.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The main study parameter is the proportion of patients with a pathological complete response (pCR) and those patients who started a wait and see strategy and have sustained clinical complete response (cCR) at 1 year. | pCR is determined after surgery directly. There is a cCR in case of a sustained clinical response until at least one year after chemoradiotherapy
  The pCR is evaluated by an experienced pathologist. A pCR is defined as the absence of residual tumour cells in the complete resected specimen including all resected regional lymph nodes (ypT0N0). A cCR is defined as the absence of viable tumour tissue based on MRI, evaluated by an experienced radiologist. There is a cCR in case of a sustained clinical response at 1 year after chemoradiotherapy.

SECONDARY OUTCOMES:
3-year and 5-year local recurrence free survival. | 3 and 5 year
  ocal recurrence is confirmed by either radiological or histopathological examination. A recurrence is registered by the treating physician in the patient's medical file.
3-year and 5-year distant metastasis free survival. | 3 and 5 year
  Distant metastases may be confirmed by either radiological or histopathological examination. Data on distant metastases are registered by the treating physician in the patient's medical file.
3-year and 5-year progression free survival. | 3 and 5 year
  Progression is defined as progression of the primary tumour, local recurrence, distant metastases confirmed by radiological or histopathological examination or death. Data regarding disease progression are registered by the treating physician in the patient's medical file.
3-year and 5-year disease free survival. | 3 and 5 year
  Disease free survival is defined as no confirmed recurrence, distant metastases or death. Disease recurrence is registered by the treating physician in the patient's medical file.
3-year and 5-year overall survival. | 3 and 5 year
  Mortality is registered in the patient's medical file which is linked to the municipal personal records database.
Radiological response after induction therapy. | Directly after induction chemotherapy
  Assessment and reporting of all MRI scans is performed according to a standard operating procedure and is registered in the patient file by the radiologist.
Radiological response after chemoradiotherapy. | 6-8 weeks after chemoradiotherapy
  Assessment and reporting of all MRI scans is performed according to a standard operating procedure and is registered in the patient file by the radiologist.
Pathologic response | Directly after surgery
  The pathologic response is graded according to the Mandard grading system. The Mandard grading is registered by the pathologist in the pathology report in the patient's medical file.
Toxicity related to induction therapy. | During induction chemotherapy
  Systemic related toxicity is graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Toxicity caused by induction therapy will be scored from day one of the first cycle of induction therapy until one month after the last administration of the induction therapy and is registered in the patient's medical file by the treating medical oncologist. Only all non-hematologic NCI-CTCAE grade 3-4 and all NCI-CTCAE ≥4 are registered.
The induction therapy compliance rate. | During induction chemotherapy
  Information on completion of induction therapy is registered by the treating medical oncologist. In all patients in whom a dose reduction is required the reason for dose reduction will be recorded in the patient's medical file.
Toxicity of chemoradiotherapy. | During chemoradiotherapy
  Chemoradiotherapy related toxicity is graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Toxicity caused by chemoradiotherapy will be scored from start of radiotherapy until 3 months after the last administration of the radiotherapy and is registered in the patient's medical file by the treating radiation oncologist. Only all non-hematologic NCI-CTCAE grade 3-4 and all NCI-CTCAE ≥4 are registered.
The compliance rate related to chemoradiotherapy. | During chemoradiotherapy
  Information on completion of chemoradiotherapy is registered by the treating radiation oncologist and registered in the patient's medical file. In all patients in whom a dose reduction is required the reason for dose reduction will be recorded in the patient's medical file.
Number of patients undergoing surgery. | immediately after surgery
  This is calculated as a percentage from the total number of patients that were included.
Type of surgery, including the use of intra-operative radiotherapy. | During the surgical procedure
  Directly after surgery, information with respect to procedure related characteristics is registered in the surgical report in the patient's medical file by the operating surgeon. Data on intra-operative radiotherapy, if administered, are registered in the patient's medical file by the treating radiation oncologist.
Major surgical morbidity rate | During admission for surgery.
  Surgical complications are graded according to the Clavien-Dindo grading system. Complications will be scored up to 3 months after surgery and are registered in the patient file by the treating physician.
Generic and cancer-specific Quality of life (QoL) assessments during treatment using Quality of life Questionnaires (QLQ) | At the moment of inclusion, after 3 months and after 12 months.
  Generic and cancer-specific quality of life assessments are assessed with QLQ-C30, a 4 point scale. Higher scores correspond with a higher response level.
Generic and cancer-specific Quality of life (QoL) assessments during treatment | At the moment of inclusion, after 3 months and after 12 months.
  Generic and cancer-specific quality of life assessments are assessed with QLQ-CR29, a 4 point scale. Higher scores represent better functioning on functional scales and a higher level of symptoms on the symptom scale.
Generic and cancer-specific Quality of life (QoL) assessments during treatment | At the moment of inclusion, after 3 months and after 12 months.
  Generic and cancer-specific quality of life assessments are assessed with EQ-5D-5L, a 5 point scale. Higher scores corresponds with a higher level of symptoms on the symptom scale.
Costs | At the moment of inclusion, after 3 months and after 12 months.
  For the purpose of economic evaluation, the EQ-5D-5L questionnaire is used at inclusion and at 3 and 12 months post-operatively. The questionnaires will be sent either by mail or digitally, according to the patient's preference.

CONTACTS AND LOCATIONS:
Overall Officials: Pim J.W.A. Burger, MD. PhD., Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (7):
- Netherlands (7):
  - Catharina Hospital Eindhoven, Eindhoven, North Brabant
  - Netherlands Cancer Institute, Amsterdam, North Holland
  - Maastricht University Medical Centre, Maastricht
  - Radboud University Medical Centre, Nijmegen
  - Erasmus MC Cancer institute, Rotterdam
  - University Medical Centre, Utrecht
  - Isala hospital, Zwolle

REFERENCES:
- [Derived] van den Berg K, Schaap DP, Voogt ELK, Buffart TE, Verheul HMW, de Groot JWB, Verhoef C, Melenhorst J, Roodhart JML, de Wilt JHW, van Westreenen HL, Aalbers AGJ, van 't Veer M, Marijnen CAM, Vincent J, Simkens LHJ, Peters NAJB, Berbee M, Werter IM, Snaebjornsson P, Peulen HMU, van Lijnschoten IG, Roef MJ, Nieuwenhuijzen GAP, Bloemen JG, Willems JMWE, Creemers GJM, Nederend J, Rutten HJT, Burger JWA. Neoadjuvant FOLFOXIRI prior to chemoradiotherapy for high-risk ("ugly") locally advanced rectal cancer: study protocol of a single-arm, multicentre, open-label, phase II trial (MEND-IT). BMC Cancer. 2022 Sep 6;22(1):957. doi: 10.1186/s12885-022-09947-w. PMID 36068495